CLINICAL TRIAL: NCT06544421
Title: The Effect of Chatbot-Assisted Nursing Education on Perceived Care Burden and Caregiver Stress
Brief Title: The Impact of Chatbot-Assisted Nursing Education on Perceived Burden of Care and Caregiver Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Esra Yılmaz Bayrakçeken, Esra Yılmaz Bayrakçeken, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: esrabayrakceken1
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chatbot; Anxiety; Depression; Stress; Caregivers
Keywords: stress; Chatbot; paralysis; Caring giver; Nursing Education; Home Care
MeSH Terms: conditions — Anxiety Disorders; Depression; Paralysis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 1 week : What is Stroke, Taking Care of the Individual with Physical Needs-1 (Experimental): Session 1 What is Stroke, The Importance of Post-Stroke Rehabilitation, Obtaining accurate health information, Contacting the Health Team, Difficult caregiving behaviors Support mechanisms in stroke patient care
  Interventions: Other: Assigned Interventions
- Week 1: What is a Stroke, Caring for Someone with Physical Needs-2 (Experimental): Session 2 Personal Care, Prevent pressure sores Position and handling techniques Pain In-bed exercises Self-care Nutrition Sleep Speech & Communication Medication Management Emotional and Cognitive Changes in the Stroke Individual
  Interventions: Other: Assigned Interventions
- Week 2: Stress of Care, Becoming resistant to stress Coping with stress-1 (Experimental): Session 1 Caregiving role barriers and facilitators Positive Aspects of Caregiving Care Stress and Its Causes, Reaction to Stress Maintaining emotional balance in the caregiving process
  Interventions: Other: Assigned Interventions
- Week 2: Stress of Care, Becoming resistant to stress Coping with stress-2 (Experimental): Self-knowledge and motivation Maintenance and Time Management Controlling the Body in the Caregiving Process Breathing and relaxation
  Interventions: Other: Assigned Interventions
- Week 3: Supporting oneself in the caregiving process and becoming resistant to stress-1 (Experimental): Session 1:
  Personal space and comfort in the care process Taking time for yourself Unreasonable beliefs and mental regulation technique Tackling anxieties
  Interventions: Other: Assigned Interventions
- Week 3: Supporting oneself in the caregiving process and becoming resistant to stress-2 (Experimental): The importance of nutrition The importance of physical activity Regulation of sleep
  Interventions: Other: Assigned Interventions
- 4 week: Control of emotions and spirituality in the process of care-1 (Experimental): Anger management Unleashing emotions and social relationships Use of humor
  Interventions: Other: Assigned Interventions
- 4 week: Control of emotions and spirituality in the process of care-2 (Experimental): Communication and Empathy Spirituality and religious coping Pray Be happy
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — Assigned Interventions

SUMMARY:
Caregivers play a key role in the provision of day-to-day care and the coordination of care services. Caregivers of stroke patients use dysfunctional coping strategies to cope with the stressors and burden of care they encounter during this long caregiving process. In this study, it will be tried to improve the stress coping skills of caregivers by using an application with chatbot support based on the COM-B model.In the study, introductory information form, stress coping styles scale, depression, anxiety, stress (DASS 21) and burden of care measurement tool will be used. The study will be conducted in a randomized controlled manner. Chatbot will be applied to the experimental group and the control group will be exposed to routine practice. The study group will consist of individuals who care for those who are discharged home from Atatürk University stroke center. Experiments and controls will be accessed by searching the hospital records. The fact that nursing education is given through a chatbot and that the chatbot is designed according to a stress training model (behavior change wheel) reflects the originality of the study. With this study, caregivers are expected to be able to manage stress effectively by teaching them how to cope with stress.

DETAILED DESCRIPTION:
gree relatives who care for the patients who receive 3-5 points from the Modified Rankin Scale will be discharged from the stroke center of the Neurology Clinic of Atatürk University Health Research and Application Center located in the city center of Erzurum.With the expectation of a 50 percent reduction in the rate of stressed patients in the intervention group and a 10 percent decrease in the control group, it was decided to include 31 people in each group with 90 percent power and 5 percent type 1 error. The sample calculation was calculated using the open epi version 3.01 web interface.It is expected that the implementation and reporting of the research will take 2 years. Year 1 Preparation of chatbot and determination of experimental controls. Implementation of training. Collection of results and writing of the report in 1 year.

The caregivers included in the experimental group will be told about the study and their written consent will be obtained. Individuals in the experimental group will be asked to apply the data collection forms prepared before the use of the application is explained. After the pre-test data is collected, a chatbot-supported application will be installed on the caregivers in the experimental group. In order for them to participate in the sessions and complete the trainings in the determined plan flow, caregivers will be called by phone and reminders will be made and checked. The sessions are expected to end in 4 weeks (8 sessions) (Gabrielli et al., 2021).A participant will be scheduled to finish the application within a maximum of 4 weeks. No intervention will be applied to the control group, they will be followed up within the scope of the routine follow-up and treatment protocol of the clinic. The chatbot-supported application, which will be prepared for stroke patient care providers, has been prepared in line with the literature using the COM-B model according to the needs of caregivers. The prepared training content was sent to the experts and the final shape was given by taking the opinions of the experts

ELIGIBILITY:
Inclusion Criteria:

* To be at least a primary school graduate
* Caregivers have the cognitive capacity to use chatbots (The chatbot application will be installed on the caregiver's android phone and the status of using it will be evaluated)
* Willingness to participate in the study
* To be open to communication and cooperation
* Having a phone with Android operating system
* Have literacy skills
* Not having participated in stress training before

Exclusion Criteria:

* Having received any psychiatric diagnosis.
* Taking antipsychotic medication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
İntroductory form | [Time Frame: up to 1 day]
  Consists of questions such as age, gender, marital status, educational status, family type, social security, occupation, having any systemic disease, duration of living with the individual care, and the status of receiving home care services.

SECONDARY OUTCOMES:
Burden of Care Scale (BVS) | [Time Frame: up to 5 week ]
  The burden of care was developed in 1980 by Zarit, Reever, and Bach-Peterson. It is a measurement tool used to evaluate the stress experienced by caregivers of individuals in need of care or the elderly. There are 22 items in the measuring tool. Substances are evaluated in Likert type.
Lazarus Coping Skills Scale | [Time Frame: up to 5 week ]
  The Lazarus Stress Coping Skills Scale is a measurement tool used to evaluate individuals' coping mechanisms with stress. Şahin and Durak (1995) developed the 30-item Stress Coping Styles Scale based on the Ways of Coping Inventory developed by Folkman and Lazarus (1985).
Depression-Anxiety-Stress (DAS-21) Scale | [Time Frame: up to 5 week ]
  DASS-21 was created by Lovibond and Lovibond by abbreviation of DAS-42 (Lovibond & Lovibond, 1995; Lovibond, 1995). The psychometric properties of the Turkish version of the "Depression, Anxiety, Stress-21" (DAS-21) scale in the normal and clinical sample were made by Sarıçam (Sarıçam, 2018).

IPD SHARING:
Plan to Share IPD: No